CLINICAL TRIAL: NCT00819949
Title: Effect of Robot-assisted Gait Training on Freezing of Gait in Parkinson's Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: B4125-K
Record Dates: First submitted 2009-01-07; First posted 2009-01-09 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2013-09

CONDITIONS: Parkinson's Disease
Keywords: Robot; Treadmill; Rehabilitation; Freezing of gait
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm 1 (Experimental): Potential eligible subjects for the trial will be individuals between ages 18-85, with a confirmed diagnosis of PD that experience freezing.
  Interventions: Device: Lokomat

INTERVENTIONS:
Device: Lokomat — The Lokomat is a motor driven exoskeleton device that employs a body weight support suspension system and treadmill. Attached to the lower limbs, the Lokomat moves the subject's legs through position controlled trajectories that mimic normal human gait patterns. This is accomplished by utilizing high quality computer-controlled motors that are precisely synchronized with the speed of the treadmill. The hip and knee joint angles are controlled in real time by software to achieve kinematically correct stepping behaviors. Each of the four motor-driven joints is individually controlled to correspond precisely to the desired joint angle trajectories. This system assures a precise match between the speed of the limb trajectory and the treadmill. In addition, sensors in the motors provide an indirect indicator of the amount of effort the patient is generating to achieve walking in an upright posture.

SUMMARY:
Freezing of gait (FOG) is a common yet poorly understood motor symptom in persons with Parkinson's disease (PD). Previous studies have shown that bilateral uncoordinated gait and gait asymmetry are related to FOG, and that intensive treadmill training in PD patients can improve gait. However, no group has yet studied the effect of robot-assisted gait training (RAGT) on FOG. The primary aim of this study is to collect pilot data on the effect of robot-assisted gait training in reducing episodes of freezing in PD.

Subjects with Parkinson's disease that experience freezing of gait will be recruited and enrolled following informed consent and screening for eligibility. Each of the 10 training session will last approximately one hour. Neurological evaluations, testing of gait parameters, and quality of life assessments will be conducted. Participants will also be asked to return for 1- and 3-month post-intervention assessments to see if the training has any lasting effects. Approximately 10-20 subjects will be enrolled, and the study will last up to 6 months.

Robot-assisted gait training will be conducted with the Lokomat (a treadmill with supplemental robot-assistance for moving the hip and knee). We will monitor changes in freezing by conducting various assessments.

There are approximately 1 million Americans with PD in the US. PD is a significant cause for reduced functional ability and quality of life, progressive disability. Patients with PD with FOG have indicated that this is one of their most disturbing symptoms, as there are no effective treatments. Therefore it is important that additional and alternative interventions for FOG be tested and developed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic PD by UK Brain Bank criteria, without other significant neurological problems.
* Men and women between the ages of 18-85 years.
* History of FOG by self-report and verified by MD.
* Must be able to walk unassisted when not freezing but use of a device to prevent falls and overcome freezing is not exclusionary. (Device should not be used for visual cueing).

Exclusion Criteria:

* Cognitively unable to understand instructions required by the study.
* Presence of medical or neurological infirmity that might contribute to significant gait dysfunction (such as severe OA, foot drop, sensory neuropathy, blindness, joint replacement, etc.), determined by the physician during the screening exam.
* Cardiovascular: recent MI < 4 wk, uncontrolled HTN >190/110 mmHg.
* History of uncontrolled diabetes.
* Significant symptoms of orthostasis when standing up.
* Circulatory problems, history of vascular claudication or 3+ pitting edema.
* Body weight over 100 kg.
* Lower extremity injuries that limit range of motion or function.
* Joint problems (hip or leg) that limit range of motion or cause pain with movement despite treatment.
* Unstable fractures.
* Pressure sores with any skin breakdown in areas in contact with the body harness or Lokomat apparatus.
* Chronic and ongoing alcohol or drug abuse.
* Active depression, anxiety or psychosis that might interfere with use of the equipment or testing.
* Inability to participate in and complete the training sessions.
* Patients determined to have an atypical parkinsonian syndrome by a neurologist.
* Patients with PD that have undergone deep brain stimulation.
* Primarily wheelchair bound.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2008-10; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Freezing of Gait | Each Visit
  Temporary halting of gait

CONTACTS AND LOCATIONS:
Overall Officials: Albert Lo, MD PhD, Principal Investigator — Providence VA Medical Center
Locations (1):
- Providence VA Medical Center, Providence, Rhode Island, United States

REFERENCES:
- [Result] Lo AC, Chang VC, Gianfrancesco MA, Friedman JH, Patterson TS, Benedicto DF. Reduction of freezing of gait in Parkinson's disease by repetitive robot-assisted treadmill training: a pilot study. J Neuroeng Rehabil. 2010 Oct 14;7:51. doi: 10.1186/1743-0003-7-51. PMID 20946640